CLINICAL TRIAL: NCT07034885
Title: Effects of Mindfulness-Based Self-Efficacy Development Program on Menopausal Symptoms and Quality of Life in Postmenopausal Women: A Randomized Controlled Trial
Brief Title: Effects of Mindfulness-Based Self-Efficacy Development Program on Postmenopausal Women
Acronym: MOPKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nurcan Gökgöz (Other Government)
Responsible Party: Sponsor-Investigator, Nurcan Gökgöz, nurse, Lokman Hekim University
Organization: Lokman Hekim University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LokmanHekimU
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Postmenopausal Period; Menopausal Symptoms; Quality of Life; Stress Management; Self-Efficacy
Keywords: Menopause; Self-Efficacy; Quality of Life; Mindfulness

STUDY DESIGN:
Intervention Model Description: This study is conducted with a randomized controlled, parallel group intervention model. Participants were divided into two groups, intervention and control groups, by simple randomization. The intervention group will be administered an 8-week Mindfulness-Based Self-Efficacy Development Program. The control group will not receive any intervention. Data from both groups will be collected with the same measurement tools before the program, at the end of the program (week 8), and 4 weeks after the end of the program.
Masking Description: In this study, blinding could not be done due to the nature of the study. Since the intervention program will be carried out directly by the researcher, the participants and the researcher will know which group is the intervention and which is the control group. However, in order to ensure impartiality in the data analysis process, the obtained data will be coded (Group 1-Group 2) and forwarded to an independent statistician and the statistical analyses will be performed by this expert without knowing the groups. Thus, it was aimed to prevent biases that may occur during the analysis phase by blinding the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the Mindfulness-Based Self-Efficacy Development Program, it is planned that the training groups will consist of a maximum of 10 people.
  The trainings will be structured as 90-120 minute sessions, 1 day a week, for a total of 8 weeks. Each session will be carried out through face-to-face training.
  The program content is structured based on Kabat-Zinn's Mindfulness-Based Stress Reduction (MBSR) protocol. The program focuses on breath awareness, focusing on bodily sensations, moving with awareness, eating with awareness and mindfulness in daily activities, coping with thoughts, emotions and stressful situations with awareness, and the present moment as a safe space within the framework of the basic components of self-compassion, intention and attitude.
  Each session will include story content appropriate to the main theme of the session. The trainings applied to the intervention group were prepared within the scope of the "Mindfulness-Based Self-Efficacy Development Program" and the co
  Interventions: Behavioral: Mindfulness-Based Self-Efficacy Development Program
- Control Group (No Intervention): The participants in the control group will be administered the measurement tools applied to the intervention group at the beginning of the study. At the end of the 8-week follow-up period, the same scales applied in the pre-test will be re-administered and interim test data will be collected. Thus, the level of change in the control group will be evaluated comparatively with the intervention group. Following the completion of the 4-week home practice applications of the intervention group, post-test data will be collected from the control group. No intervention will be applied to the participants in the control group during the study. However, in accordance with ethical principles, the content program of the sixth week of the eight-week mindfulness training applied to the intervention group will be presented to the women in the control group after the study is completed. In addition, training brochures shared with the intervention group will be provided.

INTERVENTIONS:
Behavioral: Mindfulness-Based Self-Efficacy Development Program — "Mindfulness-Based Self-Efficacy Development Program" is a unique intervention model that integrates mindfulness-based practices with self-efficacy theory, structured for postmenopausal women. With the implementation of this research, a holistic and evidence-based intervention model will be presented for physical, psychological and social problems frequently encountered in the postmenopausal period. This program processes mindfulness-based skills such as observing thoughts, body awareness, regulating emotions, coping with stress and developing self-compassion in the axis of self-efficacy development with 8-week structured sessions. In this context, it is anticipated that the study will contribute to scientific knowledge and practices.
  In addition, the "Mindfulness-Based Self-Efficacy Development Program" developed in the study aims not only at symptom management, but also at increasing the individual's perception of control over their own lives, recognizing their internal resources and
  Arms: Intervention Group

SUMMARY:
The aim of this randomized controlled clinical trial is to evaluate the effects of a mindfulness-based self-efficacy development program on menopausal symptoms and quality of life in postmenopausal women. The main questions it aims to answer are:

Does the mindfulness-based program reduce the severity of menopausal symptoms?

Does the mindfulness-based program improve the quality of life of postmenopausal women?

Does the mindfulness-based program significantly increase participants' overall self-efficacy?

The researchers will compare whether there are differences between the mindfulness-based training program applied to the intervention group and the control group in terms of menopausal symptoms, quality of life, and self-efficacy scores.

The main tasks that will be asked of the participants are as follows:

Those in the intervention group will participate in a face-to-face mindfulness-based self-efficacy development program, each session lasting at least 120 minutes, once a week for 8 weeks, with a maximum of 10 people per group.

The control group will not receive any intervention.

Participants in both groups will be evaluated with a personal information form and measurement tools such as the Menopause Symptoms Assessment Scale, the Menopause Specific Quality of Life Scale, and the General Self-efficacy Scale.

DETAILED DESCRIPTION:
This research is a randomized controlled experimental study aiming to evaluate the effects of a mindfulness-based self-efficacy development program on menopausal symptoms and quality of life in women during menopause. The research will be conducted at Lokman Hekim University Etlik Hospital between September 2025 and March 2026.

Postmenopausal women who have entered menopause naturally, who do not have a physical disability that prevents them from participating in mindfulness practices, who are literate and literate in Turkish, and who have access to technology will be included in the study. Participants will be assigned to the intervention and control groups by simple randomization.

Participants in the intervention group will receive an eight-week mindfulness-based self-efficacy development training based on Kabat-Zinn's Mindfulness-Based Stress Reduction (MBSR) program. Sessions will be held face-to-face once a week for 90-120 minutes. The program consists of components such as breath awareness, focusing on bodily sensations, mindful movement, working with emotions, and present-moment awareness.

Standard scales will be applied to all participants before and after the study to assess menopausal symptoms, quality of life and general self-efficacy levels. The collected data will be compared statistically.

This study aims to be an original study to evaluate whether a mindfulness-based self-efficacy development program has the potential to help control menopausal symptoms and improve quality of life in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Individuals who are in the +1a or +1b substage of early postmenopause according to the STRAW+10 system (at least 12 months and at most 24 months have passed since their last menstrual period)
* Are proficient in reading and writing Turkish
* Are in a spouse or partner
* Have entered menopause naturally
* Do not have a physical disability such as a severe musculoskeletal disorder, neurological disease, or mobility limitation that would prevent the use of mindfulness techniques (e.g., seated meditation, breathing exercises, gentle body awareness exercises)
* Have not used MBSR techniques in the last six months
* Own a smartphone or internet-enabled device.

Exclusion Criteria:

* Those who completed the pretest data collection forms incompletely,
* Those who had any psychological disorder or experienced a traumatic event in the last two to one years,
* Those who received hormone replacement therapy during menopause,
* Those who had any gynecological cancer

Ages: 45 Years to 57 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in menopausal symptom severity | Pre-intervention, post-intervention (week 8), follow-up (week 12)
  The severity of menopausal symptoms will be measured using the Menopausal Symptoms Rating Scale. The scale covers psychological, urogenital, and somatic dimensions. The Likert-type scale, consisting of 11 items covering menopausal complaints, includes options for each item: 0: None at all, 1: Mild, 2: Moderate, 3: Severe, and 4: Very severe. The total scale score is calculated based on the scores given for each item. The minimum possible score is 0, while the maximum is 44. A higher score indicates both an increase in the severity of menopausal symptoms and a negative impact on quality of life.
Change in quality of life | Pre-intervention, post-intervention (8th week), follow-up (12th week)
  Quality of life will be assessed with the Menopause-Related Quality of Life Scale (MENQOL). The scale includes vasomotor, psychosomatic, psychological and sexual life subscales. As the scores increase, the severity of the problems experienced increases. Lower scores indicate higher quality of life.
  On the MÖYKÖ-II, each subdomain score is ranked from 0 to 6. Women are asked to answer "no" or "yes" regarding any complaints they have experienced in the past month. If the answer is "yes," the participant scores each symptom on a scale of 0-6, indicating its presence. A "none" indicates that the symptom is not experienced, a "none" indicates that the symptom is present, and scores of 1-6 indicate the severity and increasing severity of the problem. The researcher scores each item on a scale of 1 to 8, including "none" and "none." The minimum score for each item is 1, and the maximum is 8. The minimum score for the total scale is 29, and the maximum is (29X8) 232.
Change in self-efficacy level | Pre-intervention, post-intervention (8th week), follow-up (12th week)
  Women's self-efficacy perceptions will be measured using the General Self-Efficacy Scale (GSES). The GSES is a 17-item Likert-type scale with a minimum score of 17 and a maximum score of 85. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, and 17 are reverse-scored. Higher scores indicate higher self-efficacy beliefs. The scale consists of three subscales: initiation, perseverance, and persistence.

CONTACTS AND LOCATIONS:
Overall Officials: Didem Şimşek Küçükkelepçe, Assoc. Prof. Dr., Study Director — Lokman Hekim University, Institute of Health Sciences, Department of Midwifery
Locations (1):
- Lokman Hekim Univeristy, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participants' age, gender, education level, menopause process, self-efficacy scores, quality of life and symptom management data will be shared, with their identity confidential.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing will begin 6 months after the completion of the study and publication of the results.
Access Criteria: IPD data will only be accessible to researchers who have ethics committee approval, are conducting scientific research on relevant topics, and whose data use purpose has been clearly stated.